CLINICAL TRIAL: NCT00604721
Title: A Phase 2 Study of AZD6244 in Advanced or Metastatic Hepatocellular Carcinoma
Brief Title: Selumetinib in Treating Patients With Locally Advanced or Metastatic Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00247; 07-0973; 77782; MCC-07-0973; VU-VICC-GI-0726; GCRC-2625-ORC; MCC-15260; CDR0000571751; N01CM62207 (NIH); N01CM62208 (NIH); NCT00550719 (obsolete NCT alias); NCT01656291 (obsolete NCT alias)
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2013-05

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — AZD 6244

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive a single dose of selumetinib on day 1 and undergo blood collection for PK sampling pre-dose (within 30 min of dosing), 15 and 30 minutes and 1, 2, 4, 8, 12, 24 and 48 hours post-dose. Beginning 48 hours after the initial dose and continuing until day 21, patients receive oral selumetinib twice daily. Patients also undergo blood collection for PK sampling on day 15 of course 1. In all subsequent courses, patients receive selumetinib on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: selumetinib; Other: pharmacological study

INTERVENTIONS:
Drug: selumetinib — Given orally
  Other Names: ARRY-142886; AZD6244
Other: pharmacological study
  Other Names: pharmacological studies

SUMMARY:
This phase II trial is studying selumetinib to see how well it works in treating patients with locally advanced or metastatic liver cancer. Selumetinib may stop the growth of tumor cells by blocking some of the enzymes needed for their growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To ascertain the objective response rate (complete response and partial response) in patients with locally advanced or metastatic hepatocellular carcinoma treated with AZD6244 (selumetinib).

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of AZD6244 when administered to patients with hepatocellular carcinoma and mild (Child's A to compensated Child's B) liver dysfunction.

II. To describe the pharmacokinetics (PK) of AZD6244 in this patient population and compare in exploratory fashion to the established PK profile in patients with normal hepatic function.

III. To estimate the time to event functions of progression, progression-free survival (PFS), (and PFS associated with treatment), and overall survival.

IV. To explore, preliminarily, the possible correlations between baseline mitogen-activated protein kinase (MEK) activation (i.e., presence of phospho-MEK) and radiographic response or time to progression.

V. To investigate the effects of AZD6244 on MEK kinase activity in peripheral blood mononuclear cells from patients treated with this drug.

OUTLINE:

Patients receive a single dose of selumetinib on day 1 and undergo blood collection for pharmacokinetic (PK) sampling pre-dose (within 30 min of dosing), 15 and 30 minutes and 1, 2, 4, 8, 12, 24 and 48 hours post-dose. Beginning 48 hours after the initial dose and continuing until day 21, patients receive oral selumetinib twice daily. Patients also undergo blood collection for PK sampling on day 15 of course 1. In all subsequent courses, patients receive selumetinib on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Selumetinib blood concentrations are quantified by high performance liquid chromatography. Patients also undergo tumor biopsy by CT or ultrasound guidance at baseline and on day 8. Peripheral blood mononuclear cells and tumor tissue are evaluated for mitogen-activated protein kinase baseline activity and post-treatment activity.

After completion of study treatment, patients are followed periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Meets 1 of the following criteria:

  * Histologically or cytologically confirmed hepatocellular carcinoma
  * Serum alpha fetoprotein > 1000ng/dL with characteristic imaging findings coupled with the appropriate clinical scenario (i.e., chronic hepatitis and/or cirrhosis)

    * Child's A or B cirrhosis allowed

      * If Child's B cirrhosis is present, the patient may not have significant encephalopathy or ascites that requires paracentesis and must meet laboratory criteria (i.e., well-compensated Child's B)
* Metastatic disease (including any proven lymph node metastases) or localized disease not amenable to potentially curative transplant/locoregional/surgical therapy as determined by a qualified surgeon or tumor board
* Measurable disease, defined as at least one unidimensionally measurable ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* No known brain metastases
* ECOG performance status ≤ 2
* Life expectancy > 3 months
* Leukocytes ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelets ≥ 75,000/mm³
* Total bilirubin < 2 times upper limit of normal (ULN)
* AST/ALT < 5 times ULN
* Creatinine < 1.5 mg/dL or creatinine clearance ≥ 60 mL/min
* INR < 1.4
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception before, during, and for 4 weeks after completion of study treatment
* Willing to undergo protocol-required tumor biopsies (patients must also be able to have any anticoagulation held for an appropriate period of time)
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to AZD6244 or its excipient Captisol®
* No refractory nausea and vomiting or chronic gastrointestinal diseases (e.g., inflammatory bowel disease) that would preclude adequate absorption
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* No active illicit substance or alcohol abuse
* Able to understand and willing to sign a written informed consent document
* Recovered from prior therapy
* At least 4 weeks since prior chemo embolization, radio embolization (90Y microspheres), resection, or radio frequency/cryoablation

  * Must have measurable disease outside the treated area or unequivocal evidence of disease progression within the treated area
* More than 4 weeks since prior radio therapy or major surgery
* No prior organ transplantation
* No prior systemic chemotherapy
* No prior sorafenib
* No prior therapeutic antibody or experimental systemic therapy (oral or intravenous)
* No prior hepatic artery infusion of chemotherapy
* No prior mitogen-activated protein kinase inhibitor
* No prior significant bowel resection that would preclude adequate absorption
* No concurrent fruit or juice of the grapefruit during AZD6244 therapy
* No concurrent anti retroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial agents or therapies for this cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bert O'Neil, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (6):
- United States (6):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of North Carolina, Chapel Hill, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD6244 Treatment: The first 6 patients with moderate liver dysfunction (Child's B or total bilirubin 1.5-2x ULN) were to comprise a "moderate liver dysfunction" safety cohort. AZD6244 was administered at a dose of 100 mg twice daily (48 hours after initial single dose for PK), approximately 12 hours apart, in a mix and drink formulation. For the purposes of evaluation, a cycle was defined as 21 days. Dosing for the remainder of patients (efficacy cohort) was to be determined by the algorithm presented in the safety cohort.
Period: Overall Study
Arm/Group | AZD6244 Treatment
Started | 19
Completed | 17 (2 patients failed to complete a full cycle of therapy.)
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | AZD6244 Treatment
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 4
Age, Customized [Mean (Full Range); unit: years] | 57 [48 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Radiographic Objective Response (OR)
Description: To ascertain the objective response rate (Complete Response + Partial Response [CR+PR]) of patients with the single-agent AZD6244. Our study utilized Response Evaluation Criteria in Solid Tumors (RECIST) to evaluate response.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 33 weeks
Population: Participants who completed a full 21 day cycle of therapy
Measure: Number; unit: participants
Groups:
- Safety Cohort: AZD6244 Treatment: The first 6 patients with moderate liver dysfunction (Child's B or total bilirubin 1.5-2x ULN) were to comprise a "moderate liver dysfunction" safety cohort. AZD6244 was administered at a dose of 100 mg twice daily (48 hours after initial single dose for PK), approximately 12 hours apart, in a mix and drink formulation. For the purposes of evaluation, a cycle was defined as 21 days. Dosing for the remainder of patients (efficacy cohort) was determined by the algorithm presented in the safety cohort.
Arm/Group | Safety Cohort: AZD6244 Treatment
Number analyzed (Participants) | 17
participants | 0

2. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Progression free survival has been defined as time from the start of treatment to disease progression or death as a result of any cause.
Time Frame: 33 weeks
Population: Participants who completed a full 21 day cycle of therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AZD6244 Treatment
Number analyzed (Participants) | 17
months | 1.4 [1.2 to 2.5]

3. Secondary Outcome: Median Overall Survival (OS)
Description: Overall survival has been defined as time from the start of treatment to death as a result of any cause.
Time Frame: 33 weeks
Population: Participants who completed a full 21 day cycle of therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AZD6244 Treatment
Number analyzed (Participants) | 17
months | 4.2 [1.9 to 6.0]

ADVERSE EVENTS:
Time Frame: 1 year, 5 months
Description: All 19 participants were evaluated for toxicity.
Arm/Group | AZD6244 Treatment
Serious Adverse Events (participants affected / at risk) | 8/19
Other Adverse Events (participants affected / at risk) | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD6244 Treatment (N=19)
Death - Death not associated with CTCAE term - Disease progression - 1 Event definitely related (General disorders) | 5 (5)
Hemorrhage/Bleeding - GI - Liver - Unrelated (General disorders) | 1 (1)
Hepatobiliary/Pancreas - Liver dysfunction/failure - Unrelated (Hepatobiliary disorders) | 1 (1)
Gastrointestinal - Other - Unlikely to be related (Gastrointestinal disorders) | 1 (1) — RUQ pain, nausea, dark cloudy urine - Pancreatitis
AST, SGOT - Probably related (Metabolism and nutrition disorders) | 1 (1)
AST, SGOT - Possibly related (Metabolism and nutrition disorders) | 1 (1)
Nausea - Possibly related (Gastrointestinal disorders) | 1 (1)
Hemoglobin - Possbily related (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin - Unlikely to be related (Blood and lymphatic system disorders) | 1 (1)
Bilirubin - Possibly related (Metabolism and nutrition disorders) | 1 (1)
Hemorrhage/Bleeding - GU/Urinary - Possibly related (General disorders) | 1 (1)
Fatigue - Possibly related (General disorders) | 1 (1)
Albumin, serum-low (hypoalbuminemia) - Possibly related (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was stopped at the interim analysis due to lack of radiographic response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less